CLINICAL TRIAL: NCT07276321
Title: Preliminary Efficacy of an mHealth Intervention in West Africa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Dror Ben-Zeev, Professor: School of Medicine, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00023050
Record Dates: First submitted 2025-11-18; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenic Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Treatment as Usual (No Intervention)
- FOCUS (Active Comparator)
  Interventions: Other: FOCUS
- G-FOCUS (Experimental)
  Interventions: Other: G-FOCUS

INTERVENTIONS:
Other: G-FOCUS — A cultural adaption of an evidence-based (USA populations tested) digital tool for serious mental illness
  Arms: G-FOCUS
Other: FOCUS — An evidence-based (USA populations tested) digital tool for serious mental illness.
  Arms: FOCUS

SUMMARY:
We are conducting a pilot feasibility and preliminary efficacy trial of a digital intervention for serious mental illness in West Africa.

Participants will be recruited from a large psychiatric hospital in Ghana and randomized into one of three study conditions: 1) Treatment as usual; 2) FOCUS intervention; 3) G-FOCUS intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years of age or older
2. Speaks English
3. Outpatient receiving care at Accra Psychiatric Hospital
4. Diagnosis of Schizophrenic Spectrum Disorder
5. Owns a mobile device capable of downloading smartphone applications

Exclusion Criteria:

1. Hearing, vision, or motor impairment that would hamper their ability to participate in data collection
2. Serious intellectual or developmental disability that would hamper their ability to participate in data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 6 weeks, 12 weeks
  Depressive symptoms.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline, 6 weeks, 12 weeks
  Anxiety severity
Revised Green et al Paranoid Thoughts Scale | Baseline, 6 weeks, 12 weeks
Hamilton Program for Schizophrenia Voices Questionnaire | Baseline, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dror Ben-Zeev, PhD, Principal Investigator — University of Washington
Locations (1):
- Accra Psychiatric Hospital, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No